CLINICAL TRIAL: NCT00002914
Title: PHASE II STUDY OF PIRITREXIM IN ADVANCED CARCINOMA OF THE UROTHELIUM
Brief Title: Piritrexim in Treating Patients With Advanced Cancer of the Urinary Tract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Purpose: Treatment
Other Study IDs: CDR0000065289; E-3896
Record Dates: First submitted 1999-11-01; First posted 2004-08-11 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: recurrent bladder cancer; transitional cell carcinoma of the bladder; squamous cell carcinoma of the bladder; adenocarcinoma of the bladder; recurrent urethral cancer; recurrent transitional cell cancer of the renal pelvis and ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — piritrexim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: piritrexim

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of piritrexim in treating patients with advanced cancer of the urinary tract that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the antineoplastic activity of piritrexim and its effect on the survival of patients with advanced urothelial carcinoma previously treated with systemic cytotoxic chemotherapy. II. Evaluate the toxicity of piritrexim in these patients.

OUTLINE: Patients receive piritrexim by mouth 3 times daily, 5 days a week, for 3 weeks followed by 1 week of rest. Patients with responding or stable disease continue treatment every 4 weeks until unacceptable toxicity or progression intervenes.

PROJECTED ACCRUAL: A maximum of 40 patients will be entered over 5-6 months if at least 1 response is observed in the first 14 evaluable patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed transitional cell carcinoma, squamous cell, or adenocarcinoma of the renal pelvis, ureter, bladder, or urethra Progressing regional or metastatic disease after one prior systemic or intra- arterial chemotherapy regimen Bidimensionally measurable disease, e. g.: Pulmonary nodules Palpable lymph nodes Cutaneous or subcutaneous nodules Mediastinal tumor or hepatic metastases if clearly measurable on CT No prior radiotherapy to indicator lesion unless documented progression since completion of radiotherapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0 or 1 Hematopoietic: (within 2 weeks prior to entry) WBC at least 4,000/mm3 Platelet count at least 100,000/mm3 Hepatic: (within 2 weeks prior to entry) Bilirubin no greater than 2.0 mg/dL AST no greater than twice normal Renal: (within 2 weeks prior to entry) Creatinine no greater than 1.5 mg/dL OR Creatinine clearance greater than 40 mL/min Other: No active unresolved infection No concurrent parenteral antibiotics At least 7 days since parenteral antibiotics No history of prior malignancy within 5 years except: Curatively treated nonmelanomatous skin cancer In situ cancer of the cervix Not pregnant or nursing Adequate contraception required of fertile patients Physically and medically able to take oral medications

PRIOR CONCURRENT THERAPY: Biologic therapy: One prior systemic biological response modifier therapy allowed At least 3 weeks since biologic response modifier therapy and recovered Chemotherapy: See Disease Characteristics At least 3 weeks since chemotherapy and recovered Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since radiotherapy Surgery: At least 3 weeks since major surgery and recovered

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1997-07-15 (Actual); Primary Completion 2001-06 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J. Roth, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (29):
- United States (28):
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Lakeside), Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - St. Francis Hospital/Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Roth BJ, Manola J, Dreicer R, Graham D, Wilding G; Eastern Cooperative Oncology Group. Piritrexim in advanced, refractory carcinoma of the urothelium (E3896): a phase II trial of the Eastern Cooperative Oncology Group. Invest New Drugs. 2002 Nov;20(4):425-9. doi: 10.1023/a:1020675017737. PMID 12448661